CLINICAL TRIAL: NCT01609270
Title: CardioRoot Post-Marketing Surveillance Registry
Acronym: CardioRoot
Status: Completed | Type: Observational
Sponsor: Maquet Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: MCV00008317
Record Dates: First submitted 2012-05-25; First posted 2012-05-31 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Cardiovascular Surgical Procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CardioRoot: All subjects receive the CardioRoot graft at baseline implant procedure.
  Interventions: Device: CardioRoot graft

INTERVENTIONS:
Device: CardioRoot graft — prospective single arm multi-center study to evaluate CardioRoot grafts implanted in a thoracic position.

SUMMARY:
Post-marketing surveillance registry of the CardioRoot graft.

DETAILED DESCRIPTION:
Study objective is to monitor the performance and safety of CardioRoot vascular grafts implanted in a thoracic position. Patient survival rates will be monitored as well as immediate and long-term complications.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring a CardioRoot graft as per the CardioRoot Instructions for Use (IFU)

Exclusion Criteria:

* patients with contra-indications per CardioRoot IFU
* patients requiring consecutive aortic surgery
* patients with coronary artery disease
* patients who require urgent or emergent surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with aneurysmal and occlusive disease of the thoracic aorta treated with a CARDIOROOT vascular graft.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Graft complications | 30 days
  Complications will be assessed out to one year post implantation.
Graft complications | 1 year
  Complications will be assessed out to one year post implantation.

SECONDARY OUTCOMES:
Subject mortality rate | 30 days, 1 year
  Subject mortality rate will be followed out to one year post implantation.

CONTACTS AND LOCATIONS:
Locations (6):
- Czechia (3):
  - University Hospital Olomouc, Olomouc
  - General University Hospital, Prague
  - University Hospital Motol, Prague
- Centre Hospitalier Universitaire (CHU) de Bordeaux, Bordeaux, France
- Italy (2):
  - Ospedale Manzoni di Lecco, Lecco
  - Ospedale Luigi Sacco, Milan

REFERENCES:
- [Derived] Tasca G, Lindner J, Barandon L, Santavy P, Antona C, Burkert J, Gamba A. Aortic root surgery with the CARDIOROOT vascular graft: results of a prospective multicenter post-market surveillance study. J Cardiothorac Surg. 2019 May 21;14(1):94. doi: 10.1186/s13019-019-0914-y. PMID 31113456